CLINICAL TRIAL: NCT03980717
Title: A Prospective Study on the Role of Fetal Endotracheal Occlusion (FETO) in the Resolution of Pulmonary Hypertension Among Fetuses With Severe Congenital Diaphragmatic Hernia
Brief Title: Fetal Endotracheal Occlusion (FETO) in the Resolution of Pulmonary Hypertension in Fetuses With Severe CDH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael A Belfort (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Michael A Belfort, Chairman and Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-42958
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Fetal Tracheal Occlusion; FETO plug-unplug; Goldvalve balloon; Severe Congenital Diaphragmatic Hernia; Goldbal balloon; FETO
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: The investigators will perform 40 FETO procedures on fetuses diagnosed prenatally with severe right- or left-sided CDH and outcome data will be compared with that of a control group of severe right- or left-sided CDH who will not undergo the FETO procedure because of medical or social issues. Because the prevalence of left-sided CDH is higher than right-side CDH, the investigators will perform 25 FETO procedures in left sided CDH and 15 in right-sided CDH, whose outcomes will be compared to a cohort of 40 non FETO cases. The control group will consist of patients who fit the same fetal inclusion/exclusion criteria as our FETO subjects, and will be matched by variables including maternal age, body mass index, gestational age, severity of CDH and site of CDH (left- or right-sided).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Fetal Endotracheal Occlusion (FETO) (Experimental): Placement and retrieval of the GoldBAL4 or GoldBAL2 Detachable balloon using the plug/unplug method, using BALTACCIDBPE100 Delivery Catheter.
  Interventions: Device: Goldbal Detachable Balloon and delivery microcatheter
- non-FETO (No Intervention): The control group will consist of patients who did not undergo the FETO procedure who fit the same fetal inclusion/exclusion criteria as our FETO subjects and will be matched by variables including maternal age, body mass index, gestational age, severity of CDH and site of CDH (left- or right-sided).

INTERVENTIONS:
Device: Goldbal Detachable Balloon and delivery microcatheter — Between 28+0/7 - 31+6/7 weeks gestation for severe CDH placement of the detachable balloon. Balloon retrieval will be planned for no later than 36+6/7 weeks at the discretion of the FETO center.
  Other Names: GOLDBAL4 or GOLDBAL2 Goldballoon; BALTACCIBDPE100 delivery microcatheter
  Arms: Fetal Endotracheal Occlusion (FETO)

SUMMARY:
Congenital diaphragmatic hernia (CDH) occurs when the diaphragm fails to fully fuse and leaves a portal through which abdominal structures can migrate into the thorax. In the more severe cases, the abdominal structures remain in the thoracic cavity and compromise the development of the lungs. Infants born with this defect have a decreased capacity for gas exchange; mortality rates after birth have been reported between 40-60%. Now that CDH can be accurately diagnosed by mid-gestation, a number of strategies have been developed to repair the hernia and promote lung tissue development.

Fetal tracheal occlusion (FETO), using a fetoscopically delivered and removed balloon device, has been used to temporarily occlude the trachea and increase lung distension in CDH to allow the lungs to develop and has been shown to increase survival at birth. The role of FETO in the resolution of pulmonary hypertension in fetuses with severe left- and right- sided CDH remains unclear. Our recent observation that FETO is associated with a higher proportion of infants who resolve their pulmonary hypertension by the age of 1 year as compared with those who have not had FETO, is based on a retrospective cohort study, which, as with any such design, has some intrinsic limitations. Thus, a prospective cohort study that is appropriately powered to confirm or disprove this encouraging observation is needed. If our preliminary observation is confirmed, resolution of PH by the age of 1 year could be added to the benefits of the FETO procedure in severe left and right-sided CDH cases.

The investigators will perform 40 FETO procedures on fetuses diagnosed prenatally with severe right- or left-sided CDH, and outcome data will be compared with that of a control group of severe right- or left-sided CDH who will not undergo the FETO procedure because of medical or social issues. Because the prevalence of left-sided CDH is higher than right-side CDH, the investigators will perform 25 FETO procedures in left sided CDH and 15 in right-sided CDH, and these outcomes will be compared to a cohort of 40 non FETO cases.

DETAILED DESCRIPTION:
Enrollment

Women carrying a fetus with severe CDH and a normal karyotype will undergo routine clinical evaluation. The fetus will be 28+0/7 to 31+6/7 weeks of gestational age and have severe CDH. These patients will have ultrasound and/or MRI evaluation to rule out other anomalies, calculation of the LHR from ultrasound measurements, calculation of observed/expected total lung volume and percentage of liver herniation from fetal MRI studies, echocardiography, and detailed obstetric/perinatal consultation. Patients who meet the eligibility criteria will be extensively counseled, and those who wish to participate will provide written, informed consent for the study.

Procedure

The procedure will be performed under spinal anesthesia or local anesthesia with intravenous sedation. The technique of fetal endoscopic tracheal occlusion has been described. Using standard technique, a cannula will be inserted into the amniotic cavity and a fetoscope or flexible operating endoscope will be passed through the cannula into the amniotic fluid. If, upon evaluation, the fetal trachea cannot be entered as described above, the uterus will be accessed through an incision in the belly (called a laparotomy). A laparotomy is a surgical technique tin which an incision is made in the abdomen. After the incision has been made, the uterus will be temporarily repositioned externally. The baby will then be accessed using the fetoscope and ultrasound, as described above. The laparotomy will only be performed if the baby cannot be reached and repositioned to a more favorable one by doing external maneuvers (called external version) for the FETO procedure.

The scope will be guided into the fetal larynx, and then through the fetal vocal cords with the aid of both direct vision through the scope and cross-sectional ultrasonographic visualization. A detachable latex balloon will be placed in the fetal trachea midway between the carina and the vocal cords. The balloon will be inflated with isosmotic contrast material so that it fills the fetal trachea.

Postoperative

The mothers will be discharged once stable. Serial measurements of sonographic lung volume and LHR will begin within 24-48 hours following surgery and continue weekly by targeted ultrasound evaluation. Amniotic fluid level and membrane status will also be monitored at weekly intervals. Comprehensive ultrasonography for fetal growth will be performed every four weeks (+/- 1 wk). All discharged patients will stay within 30 minutes of TCH to permit standardized postoperative management and emergent retrieval of the balloon in the event of preterm labor or premature rupture of membranes prior to the scheduled removal.

After the FETO surgery, prior to leaving the hospital, the mother will be given a medical alert bracelet identifying her as a patient with a baby with blocked airways. She will be encouraged to wear the bracelet at all times so that in case of emergency, she and others will know who to contact. She will also be given a pamphlet with instructions for medical personnel describing how to remove the balloon in case of an emergency. She should carry it with her at all times.

Balloon retrieval will be planned for no later than 36+6/7 weeks, at the discretion of the FETO center. The patient will need to commit to remaining in 30 minutes of Texas Children's Hospital Pavilion for Women until the balloon is retrieved. In the event of a patient relocating after having the balloon placed, despite having committed to remain in the area during consent process, she will be asked to return for the removal. Every effort to make arrangements for her to be managed by the nearest center capable of an EXIT procedure or balloon retrieval will be made.

After removal of the balloon, patients will have the choice of delivering at Texas Children's Hospital - Women's Pavilion with the CDH managed and repaired at TCH, or returning to their obstetrician for delivery with subsequent repair of the CDH by the pediatric surgeons at their referring facility. Given the severity of the CDH, the baby will need to be delivered in a facility that has the capability of immediate pediatric surgery services.

The investigators will need to monitor the baby at regular intervals (at 6 weeks, 3 months, 6 months, 1 year, and 2 years) after delivery to see how well the baby is breathing and how well the baby is developing. These check - ups may be at Texas Children's Hospital - Pavilion for Women or can be coordinated with doctors from the hospital of the participant's choosing.

If the child continues care at another institution, the investigators will attempt to follow up with a review of the child's medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a pregnant woman between 18 and 45 years of age
* Singleton pregnancy
* The fetuses will be 28+0/7 to 31+6/7 weeks of gestational age
* Confirmed diagnosis of severe left- or right-sided CDH of the fetus: Observed/expected total lung volume equal to or less than 0.32 with more than 21% of liver herniated into the hemithorax. (Ideally calculated between 28+0/7 and 31+6/7 weeks' gestation.)
* Normal fetal echocardiogram or echocardiogram with a minor anomaly (such a small VSD) that in the opinion of the pediatric cardiologist will not affect postnatal outcome
* Normal fetal karyotype or microarray
* The mother must be healthy enough to have surgery
* Patient and father of the baby provide signed informed consent that details the maternal and fetal risks involved with the procedure
* Patient willing to remain in Houston for the duration following balloon placement until delivery.

Exclusion Criteria:

* Contraindication to abdominal surgery, fetoscopic surgery, or general anesthesia
* Allergy to latex
* Allergy or previous adverse reaction to a study medication specified in this protocol
* Preterm labor, preeclampsia, or uterine anomaly (e.g., large fibroid tumor) in the index pregnancy.
* Fetal aneuploidy, known structural genomic variants, other major fetal anomalies that may impact the fetal/neonatal survival or known syndromic mutation
* Suspicion of major recognized syndrome (e.g. Fryns syndrome) on ultrasound or MRI
* Maternal BMI >40
* High risk for fetal hemophilia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of Pulmonary Hypertension - 6 months | by the age of 6 months
  To compare the proportion of fetuses with resolution of PH by the age of 6 months in neonates with severe CDH who underwent the FETO procedure and that of a control group composed of neonates who did not have the FETO procedure.
Resolution of Pulmonary Hypertension - 12 months | by the age of 12 months
  To compare the proportion of fetuses with resolution of PH by the age of 12 months in neonates with severe CDH who underwent the FETO procedure and that of a control group composed of neonates who did not have the FETO procedure.

SECONDARY OUTCOMES:
2-year Survival | 2 years after childbirth
  To assess two-year neonatal survival following FETO.
Number of participants who undergo a successful completion of surgical procedures/balloon placement | Up to 10 weeks
  To assess the successful completion of surgical procedures/placement of balloons in fetuses with severe CDH. Case report forms are utilized to record study related data, including any procedural complications such as failed balloon placement or failed balloon retrieval, as well as surgical or anesthesia complications. At least twice a month fetal surveillance will be performed for up to 10 weeks post balloon placement.
Maternal Outcomes- Maternal Morbidity-incidence of preterm delivery | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of preterm delivery (spontaneous or indicated).
Maternal Outcomes- Maternal Morbidity-incidence of cesarean section | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of cesarean section rate.
Maternal Outcomes- Maternal Morbidity-length of hospitalization | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of length of hospitalization after the FETO procedure.
Maternal Outcomes- Maternal Morbidity- length of hospitalization after UNPLUG procedure | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of length of hospitalization after balloon removal (UNPLUG)
Maternal Outcomes- Maternal Morbidity- vaginal bleeding | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of post procedure vaginal bleeding.
Maternal Outcomes- Maternal Morbidity- Placental abruption | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of post-procedure placental abruption.
Maternal Outcomes- Maternal Morbidity- Rupture of membranes | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of post-procedure rupture of membranes. Amniotic fluid level and membrane status will also be monitored at weekly intervals by ultrasonography.
Maternal Outcomes- Maternal Morbidity- oligohydramnios | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of post-procedure oligohydramnios.Amniotic fluid level and membrane status will also be monitored at weekly intervals by ultrasonography.
Maternal Outcomes- Maternal Morbidity- chorioamnionitis | Up to 6 weeks postpartum
  Case report forms are utilized to record study related data through patient's medical chart review. Maternal morbidity will be assessed in terms of incidence of post-procedure chorioamnionitis.
Neonatal/Child outcomes- Pulmonary Morbidity - Number of babies that require ECMO | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Short-term measures of neonatal pulmonary morbidity, including the need for extracorporeal membrane oxygenation.
Neonatal/Child outcomes- Pulmonary Morbidity- ventilatory support | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Short-term measures of neonatal pulmonary morbidity, including the duration of neonatal ventilatory support.
Neonatal/Child outcomes- Pulmonary Morbidity- Number of participants that require the use of supplemental oxygen | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Short-term measures of neonatal pulmonary morbidity, including the need for administration of supplemental oxygen.
Neonatal/Child outcomes- gastrointestinal morbidity | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Short-term measures of gastrointestinal morbidity.
Neonatal/Child outcomes-neurologic morbidity | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Short-term measures of neurologic morbidity.
Neonatal/Child outcomes- Survival to discharge from the hospital | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Survival to discharge from the hospital.
Neonatal/Child outcomes- Duration of hospitalization. | Up to 2 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Duration of hospitalization after delivery.
Neonatal/Child outcomes- Number of participants that need supplemental oxygen | Up to 18 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Assessments of measures of long-term morbidity as the need for supplemental oxygen.
Neonatal/Child outcomes- recurrent infection | Up to 18 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Assessments of measures of long-term morbidity as the rates of recurrent infection.
Neonatal/Child outcomes- repeated hospitalization | Up to 18 years of age
  Case report forms are utilized to record study related data through patient's medical chart. Assessments measures of long-term morbidity as the need for repeated hospitalization. A general health questionnaire will also be given in the form of an interview, either face to face or over the phone. The questionnaire contains questions regarding the children's health status; including hospitalizations, medications, surgical procedures, medical interventions and additional therapies he/she is receiving, and questions to evaluate his/her behavioral and social development.
Neonatal/Child outcomes- Neurodevelopmental | Up to 18 years of age
  Developmental Profile questionnaire will be utilized to record study related data. Assessments of neurodevelopmental outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belfort, MD PhD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deprest J, Jani J, Gratacos E, Vandecruys H, Naulaers G, Delgado J, Greenough A, Nicolaides K; FETO Task Group. Fetal intervention for congenital diaphragmatic hernia: the European experience. Semin Perinatol. 2005 Apr;29(2):94-103. doi: 10.1053/j.semperi.2005.04.006. PMID 16050527
- [Background] Deprest J, Jani J, Van Schoubroeck D, Cannie M, Gallot D, Dymarkowski S, Fryns JP, Naulaers G, Gratacos E, Nicolaides K. Current consequences of prenatal diagnosis of congenital diaphragmatic hernia. J Pediatr Surg. 2006 Feb;41(2):423-30. doi: 10.1016/j.jpedsurg.2005.11.036. PMID 16481263
- [Background] Done E, Gucciardo L, Van Mieghem T, Jani J, Cannie M, Van Schoubroeck D, Devlieger R, Catte LD, Klaritsch P, Mayer S, Beck V, Debeer A, Gratacos E, Nicolaides K, Deprest J. Prenatal diagnosis, prediction of outcome and in utero therapy of isolated congenital diaphragmatic hernia. Prenat Diagn. 2008 Jul;28(7):581-91. doi: 10.1002/pd.2033. PMID 18634116
- [Background] Saura L, Castanon M, Prat J, Albert A, Caceres F, Moreno J, Gratacos E. Impact of fetal intervention on postnatal management of congenital diaphragmatic hernia. Eur J Pediatr Surg. 2007 Dec;17(6):404-7. doi: 10.1055/s-2007-989275. PMID 18072025
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Kohl T, Gembruch U, Tchatcheva K, Schaible T. Current consequences of prenatal diagnosis of congenital diaphragmatic hernia by Deprest et al (J Ped Surg 2006;41:423-30). J Pediatr Surg. 2006 Jul;41(7):1344-5; author reply 1345-6. doi: 10.1016/j.jpedsurg.2006.04.001. No abstract available. PMID 16818078
- [Background] Harrison MR, Adzick NS, Estes JM, Howell LJ. A prospective study of the outcome for fetuses with diaphragmatic hernia. JAMA. 1994 Feb 2;271(5):382-4. PMID 8054005
- [Background] Style CC, Olutoye OO, Belfort MA, Ayres NA, Cruz SM, Lau PE, Shamshirsaz AA, Lee TC, Olutoye OA, Fernandes CJ, Cortes MS, Keswani SG, Espinoza J. Fetal endoscopic tracheal occlusion reduces pulmonary hypertension in severe congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2019 Dec;54(6):752-758. doi: 10.1002/uog.20216. Epub 2019 Nov 4. PMID 30640410
- [Background] Belfort MA, Olutoye OO, Cass DL, Olutoye OA, Cassady CI, Mehollin-Ray AR, Shamshirsaz AA, Cruz SM, Lee TC, Mann DG, Espinoza J, Welty SE, Fernandes CJ, Ruano R. Feasibility and Outcomes of Fetoscopic Tracheal Occlusion for Severe Left Diaphragmatic Hernia. Obstet Gynecol. 2017 Jan;129(1):20-29. doi: 10.1097/AOG.0000000000001749. PMID 27926636